CLINICAL TRIAL: NCT02085668
Title: A Prospective, Multicenter, Randomized, Open-label, Feasibility, Safety and Efficacy Study of Renal Denervation in Patients With Chronic Heart Failure (CHF)
Brief Title: Renal Denervation in Patients With Chronic Heart Failure
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: This study was stopped after the publication of the Symplicity HTN-3 trial even before patient inclusion.
  The protocol (including the renal denervation device) were revised and a new trial conducted ( NCT04947670).
Sponsor: University Hospital, Saarland (Other)
Responsible Party: Sponsor
Organization: Universität des Saarlandes (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RE-ADAPT-HF; CIV-13-10-011660 (Other: EUDAMED Number European Databank on Medical Devices)
Record Dates: First submitted 2014-03-10; First posted 2014-03-13 (Estimated); Last update posted 2023-05-26 (Actual); Status verified 2023-05

CONDITIONS: Chronic Heart Failure; Cardio-Renal Syndrome
Keywords: Chronic Heart Failure; Cardio-Renal Syndrome; Renal Denervation; Symplicity; Sympathetic activation
MeSH Terms: conditions — Cardio-Renal Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Treatment Group (Experimental): Renal denervation and maintenance of heart failure medications
  Interventions: Device: Renal denervation (Symplicity™)
- Control Group (No Intervention): Maintenance of heart failure medications with option for cross-over renal denervation treatment after 6-months

INTERVENTIONS:
Device: Renal denervation (Symplicity™) — Delivery of radiofrequency through the wall of the renal artery to disrupt the surrounding renal nerves under angiography control
  Other Names: Renal denervation with Symplicity™ Renal Denervation System
  Arms: Treatment Group

SUMMARY:
The purpose of the trial is to investigate the safety and effectiveness of renal denervation for the treatment of chronic heart failure (CHF).

DETAILED DESCRIPTION:
Heart failure is a major public health problem. It is associated with high mortality, frequent hospitalization and represents a large cost to the health care system. Therapies to ameliorate the high mortality and morbidity of heart failure have focused on abrogation of activated neurohormonal systems associated with this condition. These systems include the renin-angiotensin-aldosterone system and the sympathetic nervous system.

Strategies to ameliorate sympathetic activation have primarily focused on blockade of the beta-adrenoceptors that mediate the adverse effects of activation of this system upon the myocardium. This has been a highly successful strategy with beta-blockers resulting in an approximately 35% reduction in mortality as well as improvements in hospitalization and quality of life and attenuation of disease progression.

However, less than full blockade of the effects of the sympathetic nervous system is achieved with the use of conventional doses of beta-blockers. Moreover, a not insignificant fraction of patients are unable to tolerate beta-blockers or are not able to have them up-titrated to target effective doses, in large part because of the systemic nature of these agents, whereas renal denervation allows the selective removal of the kidney's contribution to central sympathetic drive without blunting other compensatory mechanisms.

The renin-angiotensin-aldosterone axis has also been found to be a key system involved in heart failure disease progression and it too may be inhibited by renal sympathetic denervation.

Therefore, a clear need exists for further strategies to beneficially manipulate the sympathetic activation that is characteristic of the heart failure disease process.

Cardiorenal syndrome is a major comorbid condition of patients with advanced chronic heart failure. In the setting of renal hypoperfusion and/or activation of neurohormonal and cytokine systems there is a reduction in glomerulofiltration. Renal function has been found to be a major determine of prognosis in these patients. Strategies to ameliorate cardiorenal syndrome are being actively pursued. There is considerable a priori evidence to suggest that the sympathetic nervous system, in particular renal sympathetic, is a key factor to the progression of cardiorenal syndrome and impaired tubulo-glomerular feedback. In particular renal sympathetics reduce renal perfusion through vascular alpha adrenergic receptor stimulation as well as, indirectly, through stimulation of local release of adenosine causing afferent glomerular arteriole constriction. We hypothesize that by disrupting renal sympathetic afferent and efferent activity these salutary adenosine inhibitory mediated effects will be demonstrated using the renal denervation approach.

A number of studies with hypertension patients indicate that the Symplicity Catheter System can safely denervate the kidney without significant periprocedural complications.

In a small first-in man pilot study, involving seven normotensive patients with chronic heart failure, six months after renal denervation their 6-min walk distance improved significantly and the patients' self-assessment of well-being also improved. No procedural or post procedural complications following renal denervation in patients in 6 months of intensive follow-up were found.

The investigators believe that therapeutic renal denervation using the Symplicity Catheter is a promising therapy for patients with elevated sympathetic activity, as in CHF.

ELIGIBILITY:
Inclusion Criteria:

* New York Heart Association Class II-III symptoms of chronic heart failure
* Systolic left ventricular dysfunction as assessed by echocardiogram with left ventricular ejection fraction in a range of 10%- 40%.
* GFR >30 mL/min/1.73m2
* Brain natriuretic Peptide (BNP) >100 pg/ml or N terminal (NT)-Pro-BNP >400 pg/ml.
* Optimal medical therapy according to current guidelines for CHF management. Treatment for HF must be stable (including drug and dose) for at least 4 weeks prior to procedure, with the exception of diuretics, where stability is required for at least 2 weeks.
* others

Exclusion Criteria:

* Renal arterial anatomy that is ineligible for treatment
* CHF caused by pericarditis or by acute myocarditis or by endocrine diseases.
* Myocardial infarction, unstable angina pectoris, or a cerebrovascular accident within three 12 weeks of the screening visit.
* Office systolic BP at screening less than 90 mmHg
* Primary pulmonary hypertension.
* Clinically significant cardiac structural valvular disease, unless corrected by a properly functional prosthetic valve
* Major surgery, including bariatric surgery, in the previous 12 weeks before baseline.
* Contrast media administration in the previous 30 days before baseline.
* Known hypersensitivity to material of the Symplicity Catheter.
* Inpatient hospitalization for decompensated HF in the previous 60 days before baseline.
* others

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-05; Primary Completion 2015-12 (Estimated); Study Completion 2019-05 (Estimated)

PRIMARY OUTCOMES:
Safety of renal denervation with the Symplicity Catheter System with special consideration of clinically significant periprocedural adverse events in CHF patients | Baseline visit for treatment group, month 6 visit for control group
  Number of complications associated with the delivery and/or use of the Symplicity Catheter (e.g., vascular injury and bleeding complications, access site hematoma, etc.).
  Vital signs, blood and urine measurements taken before, during and after the denervation procedure

SECONDARY OUTCOMES:
Physiologic response to renal denervation: ventricular function | From denervation prodecure to 6 months after renal denervation procedure
  Measured by echocardiography at 6 months
Physiologic Response to renal denervation: renal function | From denervation prodecure to 6 months after renal denervation procedure
  Calculated by glomerular filtration rate (GFR) at 6 months
Physiologic Response to renal denervation: symptomatology/Quality of Life | From denervation prodecure to 6 months after renal denervation procedure
  Measured by EuroQol - 5 dimensions (EQ-5D) and by Kansas City Cardiomyopathy questionnaires at 6 months after renal denervation
Physiologic Response to renal denervation: additional parameters | From denervation prodecure to 6 months after renal denervation procedure
  Composite measure

CONTACTS AND LOCATIONS:
Overall Officials: Michael Böhm, MD, Principal Investigator — University Hospital, Saarland
Locations (11):
- Paracelsus Medical University, Salzburg, Austria
- Germany (8):
  - University Heart Center Freiburg Bad Krozingen, Bad Krozingen
  - German Heart Institute Berlin, Berlin
  - University Hospital Bonn, Bonn
  - University Hospital Gießen Marburg, Giessen
  - University Hospital Heidelberg, Heidelberg
  - University Hospital Saarland, Homburg/Saar
  - University of Leipzig, Heart Center, Leipzig
  - University Hospital Tübingen, Tübingen
- Sahlgrenska University Hospital, Gothenburg, Sweden
- University Hospital Zurich, Zurich, Switzerland